CLINICAL TRIAL: NCT03208803
Title: Patients With Myelofibrosis Treated With Combination of Janus Kinase 2 Inhibitor and Erythropoiesis-stimulating Agent. A French Observational Study.
Brief Title: Combination of JAK2 Inhibitor and Erythropoiesis-stimulating Agent in Myelofibrosis
Acronym: Ruxo-EPO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Other Study IDs: 15-10_Ruxo-EPO
Record Dates: First submitted 2017-06-28; First posted 2017-07-06 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Myelofibrosis; Anemia
Keywords: Myelofibrosis; Erythropoiesis-stimulating Agents; Janus Kinase 2 inhibitors; Ruxolitinib
MeSH Terms: conditions — Primary Myelofibrosis; Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
In patients with myelofibrosis, ruxolitinib is a current therapeutic option, which has demonstrated rapid and durable reduction in splenomegaly and improved disease-related symptoms. Anemia is another frequent issue in myelofibrosis. Consistent with its JAK2 signalling inhibition, ruxolitinib therapy has been shown to be detrimental on the hemoglobin level, increasing the depth of anemia or transfusion need.

Despite potential antagonistic mechanisms of action on Janus Kinase 2, some responses on anemia have been reported with the addition of Erythropoiesis-stimulating Agent to ruxolitinib in a small subset of patients in the COMFORT II study.

Ruxo-EPO is an observational study aimed to better assess the combination of Erythropoiesis-stimulating Agent and a Janus Kinase 2 inhibitor for therapeutic efficacy on anemia, Myelofibrosis evolution and for tolerance, in a larger cohort of patients treated for myelofibrosis in general practice.

DETAILED DESCRIPTION:
Myeloproliferative Neoplasms are chronic diseases; they encompass Polycythemia Vera, Essential Thrombocythemia, and Primary Myelofibrosis with shared mutations that constitutively activate the physiologic signal-transduction pathways responsible for hematopoiesis. Myelofibroses may arise either as primary or antecedent to Polycythemia Vera and Essential Thrombocythemia. Myelofibrosis is the least common and the most aggressive of these diseases leading to death in 5 to 7 years due to bone marrow failure, massive splenomegaly related to extra medullary hematopoiesis, constitutional symptoms and cachexia.

Until recently, treatment of Myelofibrosis consisted of supportive care only, especially transfusions.

Since 2005 driver mutations have been identified in more than 90% of patients with myeloproliferative neoplasms, providing substantial insight into their pathogenesis and leading to the development of JAK inhibitor drugs. Ruxolitinib, the first one available, has shown activity whatever the presence of Janus Kinase 2 mutation, in reducing splenomegaly, improving cytopenias, alleviating constitutional symptoms and finally improving survival (COMFORT I and II studies). In France, access to ruxolitinib has been possible since April 2011, before wider availability in November 2012.

Anemia is a frequent issue in Myelofibrosis, which may be managed by the use of Erythropoiesis-stimulating Agent, leading to a 40-50% response rate in small studies.

Consistent with its Janus Kinase 2 signalling inhibition, ruxolitinib therapy has been shown to be detrimental on the hemoglobin level, increasing the depth of anemia or transfusion need, especially during the first 12-24 weeks of treatment in the COMFORT studies.

Despite potential antagonistic mechanisms of action on Janus Kinase 2, some responses on anemia have been reported with the addition of Erythropoiesis-stimulating Agent to ruxolitinib in a small subset of patients in the COMFORT II study.

Ruxo-EPO is an observational study aimed to better assess the combination of Erythropoiesis-stimulating Agent and a Janus Kinase 2 inhibitor for therapeutic efficacy on anemia, Myelofibrosis evolution and for tolerance, in a larger cohort of patients treated for myelofibrosis in general practice.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary myelofibrosis or post-polycythemia myelofibrosis or post-essential thrombocythemia myelofibrosis
* previously started with a combination of Janus Kinase 2 Inhibitor and Erythropoiesis-stimulating Agent, whatever the date during the course of their disease

Exclusion Criteria:

- patients who denied participating to this observational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myelofibroses treated with a combination of Janus Kinase 2 Inhibitor and Erythropoiesis-stimulating Agent in one of the France Intergroup Myeloproliferative neoplasms centers
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Effect on anemia of the combination Janus Kinase 2 Inhibitor and Erythropoiesis-stimulating Agent | 6 months
  Response rate assessed with 2006 International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) and European Leukemia Network (ELN) criteria

SECONDARY OUTCOMES:
Patterns of the combination Janus Kinase 2 Inhibitor and Erythropoiesis-stimulating Agent | 6 months
  Modalities of the combination (drugs of interest begun at the same or at different dates, order of the drug combination if started at different dates, duration of combination, doses of each drug)
Patients and Myelofibrosis characteristics | at inclusion
  Demographic characteristics of included patients, Characteristics of diseases (date of diagnosis, primary or secondary myelofibrosis, prognostic scores, level of hemoglobin, transfusion dependency, splenomegaly, mutations, delay between myelofibrosis diagnosis and Jak2 inhibitor treatment)
Response rate of the combination treatment on constitutional symptoms of myelofibrosis | 3 years
Response rate of the combination treatment on splenomegaly | 3 years
  Splenomegaly size assessment
Efficacy of the combination treatment on bone marrow fibrosis | 3 years
  Assessment of bone marrow fibrosis change if bone marrow biopsy has been done
Efficacy of the combination treatment on Janus Kinase 2 allelic burden change | 3 years
  Assessment of Janus Kinase 2 allelic burden change if molecular evaluation has been done in blood
Adverse Events on combination treatment | 3 years
Overall survival on combination treatment | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Malak, MD, Principal Investigator — Hôpital René Huguenin - Institut Curie - St Cloud - France; Lydia Roy, MD, Study Director — Hôpital Henri Mondor - Créteil - France; Pascale Cony-Makhoul, MD, Study Director — CH Annecy Genevois - Pringy - France; Mathieu Wemeau, MD, Study Director — CH Arras

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cervantes F. How I treat myelofibrosis. Blood. 2014 Oct 23;124(17):2635-42. doi: 10.1182/blood-2014-07-575373. Epub 2014 Sep 16. PMID 25232060
- [Background] James C, Ugo V, Le Couedic JP, Staerk J, Delhommeau F, Lacout C, Garcon L, Raslova H, Berger R, Bennaceur-Griscelli A, Villeval JL, Constantinescu SN, Casadevall N, Vainchenker W. A unique clonal JAK2 mutation leading to constitutive signalling causes polycythaemia vera. Nature. 2005 Apr 28;434(7037):1144-8. doi: 10.1038/nature03546. PMID 15793561
- [Background] Verstovsek S, Mesa RA, Gotlib J, Levy RS, Gupta V, DiPersio JF, Catalano JV, Deininger MW, Miller CB, Silver RT, Talpaz M, Winton EF, Harvey JH Jr, Arcasoy MO, Hexner EO, Lyons RM, Raza A, Vaddi K, Sun W, Peng W, Sandor V, Kantarjian H; COMFORT-I investigators. Efficacy, safety, and survival with ruxolitinib in patients with myelofibrosis: results of a median 3-year follow-up of COMFORT-I. Haematologica. 2015 Apr;100(4):479-88. doi: 10.3324/haematol.2014.115840. Epub 2015 Jan 23. PMID 25616577
- [Background] Cervantes F, Vannucchi AM, Kiladjian JJ, Al-Ali HK, Sirulnik A, Stalbovskaya V, McQuitty M, Hunter DS, Levy RS, Passamonti F, Barbui T, Barosi G, Harrison CN, Knoops L, Gisslinger H; COMFORT-II investigators. Three-year efficacy, safety, and survival findings from COMFORT-II, a phase 3 study comparing ruxolitinib with best available therapy for myelofibrosis. Blood. 2013 Dec 12;122(25):4047-53. doi: 10.1182/blood-2013-02-485888. Epub 2013 Oct 30. PMID 24174625
- [Background] Ellis MH, Lavi N, Mishchenko E, Dally N, Lavie D, Courevitch A, Gutwein O, Bulvik S, Braester A, Chubar E, Tavor S, Duek A, Kirgner I, Koren-Michowitz M. Ruxolitinib treatment for myelofibrosis: Efficacy and tolerability in routine practice. Leuk Res. 2015 Aug 12:S0145-2126(15)30356-8. doi: 10.1016/j.leukres.2015.08.003. Online ahead of print. PMID 26364797
- [Background] McMullin MF, Harrison CN, Niederwieser D, Demuynck H, Jakel N, Gopalakrishna P, McQuitty M, Stalbovskaya V, Recher C, Theunissen K, Gisslinger H, Kiladjian JJ, Al-Ali HK. The use of erythropoiesis-stimulating agents with ruxolitinib in patients with myelofibrosis in COMFORT-II: an open-label, phase 3 study assessing efficacy and safety of ruxolitinib versus best available therapy in the treatment of myelofibrosis. Exp Hematol Oncol. 2015 Sep 15;4:26. doi: 10.1186/s40164-015-0021-2. eCollection 2015. PMID 26380150
- [Background] Tefferi A, Cervantes F, Mesa R, Passamonti F, Verstovsek S, Vannucchi AM, Gotlib J, Dupriez B, Pardanani A, Harrison C, Hoffman R, Gisslinger H, Kroger N, Thiele J, Barbui T, Barosi G. Revised response criteria for myelofibrosis: International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) and European LeukemiaNet (ELN) consensus report. Blood. 2013 Aug 22;122(8):1395-8. doi: 10.1182/blood-2013-03-488098. Epub 2013 Jul 9. PMID 23838352